CLINICAL TRIAL: NCT06105242
Title: Biological Sex and Sex Hormones Moderate Right Ventricular (RV) Dysfunction and Recovery in Chronic Thromboembolic Pulmonary Hypertension
Brief Title: Biological Sex and CTEPH-related RV Dysfunction and Recovery (BIOSPHeRe)
Status: Recruiting | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1051738
Record Dates: First submitted 2022-10-17; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: CTEPH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective Cohort Aim 1: Aims 1 and 2 are retrospective and will be conducted with the same dataset, just at two different time points (at diagnosis of CTEPH and after PTE surgery). For simplicity, aims 1 and 2 will be combined into one section throughout the protocol.
- Retrospective Cohort Aim 2: Aims 1 and 2 are retrospective and will be conducted with the same dataset, just at two different time points (at diagnosis of CTEPH and after PTE surgery). For simplicity, aims 1 and 2 will be combined into one section throughout the protocol.
- Prospective Cohort Aim 3: Aim 3 is prospective and will enroll a distinct set of patients from Aim 1 and 2.

SUMMARY:
1. To identify biological sex differences in baseline RV function in CTEPH
2. To identify biological sex differences in recovery of RV function after PTE surgery in CTEPH
3. To determine if sex hormone levels relate to RV function at CTEPH diagnosis and during recovery after PTE.

DETAILED DESCRIPTION:
Aims 1 and 2 together comprise a retrospective cohort study. We will identify historical subjects with newly diagnosed CTEPH using a clinical database. We will perform TTE strain analysis (RVGLS) to compare RV function between the biologic sexes at diagnosis and after surgical correction of CTEPH (to assess recovery).

ELIGIBILITY:
Inclusion criteria

* Adult (≥18 years old) patients diagnosed with CTEPH per current guideline standard42
* Subject must have a baseline TTE (within 3 months of diagnosis) with adequate images for RVGLS analysis
* Subject must have a right heart catheterization (RHC) at the time of diagnosis
* To be included in the Aim 2 analysis, patients must undergo PTE surgery and have a TTE performed 3-9 months after surgery with adequate images for RVGLS strain analysis

Exclusion criteria

* Unclear or mixed PH diagnosis as designated by an expert clinician at Intermountain PH center
* Any subjects <18 years of age
* Patients diagnosed during pregnancy
* Patients without a TTE and RHC at time of diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with right ventricular failure
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Biosphere | 1 year
  To assess biological sex differences in baseline RV function in CTEPH
Biopshere | 1 year
  To determine the biological sex differences in recovery of RV function after PTE surgery in CTEPH
Biosphere | 1 year
  To assess if and how sex hormone levels relate to RV function at CTEPH diagnosis and during recovery after PTE.

CONTACTS AND LOCATIONS:
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided